CLINICAL TRIAL: NCT06824168
Title: A Phase 2, Multicenter, Randomized, Open-label Trial to Evaluate Safety and Efficacy of Two Dose Levels of Quizartinib as Maintenance for Adult Patients With Newly Diagnosed FLT3-ITD (+) Acute Myeloid Leukemia in Complete Remission
Brief Title: Evaluation of Two Dose Levels of Quizartinib as Maintenance in FLT3-ITD (+) Acute Myeloid Leukemia Patients in Complete Remission
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AC220-167
Record Dates: First submitted 2025-02-07; First posted 2025-02-13 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Acute Myeloid Leukemia; Leukemia
Keywords: acute myeloid leukemia; quizartinib; FLT3; allo-HSCT; leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia | interventions — quizartinib

STUDY DESIGN:
Masking Description: This is an open-label study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): Participants will receive higher dose of quizartinib
  Interventions: Drug: Quizartinib High Dose
- Arm 2 (Experimental): Participants will receive lower dose of quizartinib
  Interventions: Drug: Quizartinib Low Dose

INTERVENTIONS:
Drug: Quizartinib High Dose — Participants in Arm 1 will receive oral daily higher dose of quizartinib,
  Other Names: VANFLYTA®
  Arms: Arm 1
Drug: Quizartinib Low Dose — Participants in Arm 2 will receive oral daily lower dose of quizartinib
  Other Names: VANFLYTA®
  Arms: Arm 2

SUMMARY:
This clinical two-arm trial is designed to evaluate two doses of quizartinib as maintenance therapy after induction/consolidation in participants with FMS-like tyrosine kinase 3 (FLT3)-internal tandem duplication (ITD) (+) acute myeloid leukemia (AML) in first complete remission (CR) who have not received allogeneic hematopoietic stem cell transplantation (allo-HSCT).

DETAILED DESCRIPTION:
This study also involves the Holter sub-study, which is designed to assess the impact of rapid acceleration in heart rate on the cardiac safety of quizartinib.

ELIGIBILITY:
Key Inclusion Criteria:

1. Adults ≥18 years of age or the minimum legal adult age (whichever is greater) on the day of signing the ICF (no upper limit of age).
2. Newly diagnosed, morphologically documented primary AML or AML secondary to myelodysplastic syndrome or a myeloproliferative neoplasm based on the World Health Organization (WHO) 2008/2016 classification.
3. Participant has confirmed FLT3-ITD-positive (≥0.05 SR or ≥5% VAF) activating mutation from initial diagnosis in bone marrow or peripheral blood as determined by a local institution's validated molecular testing.
4. Participants must have confirmed, morphologically documented CR1, on the most recent BMA, based on the local laboratory results, performed within 28 days prior to C1D1 of maintenance therapy. Complete remission will be defined as <5% blasts in the bone marrow with no morphologic characteristics of acute leukemia (e.g., Auer Rods), no evidence of extramedullary disease, and no leukemic blasts in the peripheral blood.

   Complete blood count recovery is required with absolute neutrophil count of more than 1.000 × 109/L and platelets more than 100 × 109/L (IWG criteria).27
5. Participant must meet the following prior therapy requirements:

   1. Has received at least one cycle of induction therapy but no more than two to achieve CR1. The induction cycles can be the same regimen or different regimens and may contain conventional agents only (e.g., cytarabine + daunorubicin or idarubicin: "7 + 3" or "5 + 2"), or a combination with FLT3 inhibitors.
   2. Has not received more than four cycles of consolidation therapy. Regimens may contain conventional agents only.
   3. FLT3 inhibitors are permitted as part of the induction or consolidation treatment.

   Participants who received FLT3 inhibitors before enrollment in the trial will need a washout period of 14 days.
6. Able to begin the maintenance phase within 60 days of D1 of the last consolidation cycle received.
7. Eastern Cooperative Oncology Group (ECOG) PS of 0 to 2.

Key Exclusion Criteria:

1. Diagnosis of acute promyelocytic leukemia (APL), French-American-British classification M3 or WHO classification of APL with translocation, t(15;17)(q22;q12), or BCR-ABL positive leukemia (i.e., chronic myelogenous leukemia in blast crisis); participants who undergo diagnostic workup for APL and treatment with all-trans retinoic acid (ATRA), but who are found not to have APL, are eligible (treatment with ATRA must be discontinued before starting induction chemotherapy).
2. Diagnosis of AML secondary to prior chemotherapy or radiotherapy for other neoplasms.
3. Prior treatment for AML, except for the following allowances:

   1. Induction and consolidation therapy, as previously described (inclusion criterion #5)
   2. Leukapheresis
   3. Hydroxyurea to treat hyperleukocytosis
   4. Cranial radiotherapy for central nervous system (CNS) leukostasis
   5. Prophylactic intrathecal chemotherapy
   6. Growth factor/cytokine support
4. Participant had received allo-HSCT as part of AML treatment.
5. Treatment with any strong or moderate CYP3A inducers within 2 weeks or 5 half-lives of randomization whichever is longer
6. Uncontrolled or significant cardiovascular disease, including the following:

   1. QTcF interval >450 ms (based on average of triplicate ECG at Screening)
   2. Diagnosed or suspected congenital long QT syndrome or known family history of congenital long QT syndrome
   3. History of clinically relevant ventricular arrhythmias, such as ventricular tachycardia, ventricular fibrillation, or Torsade de Pointes
   4. Participant has bradycardia of less than 50 beats per minute (bpm; as determined by central reading), unless the participant has a pacemaker
   5. History of second- or third-degree heart block. Candidates with a history of heart block may be eligible if they currently have pacemakers and have no history of fainting or clinically relevant arrhythmia with pacemakers.
   6. Myocardial infarction within 6 months prior to screening
   7. Uncontrolled angina pectoris within 6 months prior to screening
   8. New York Heart Association Class 3 or 4 congestive heart failure
   9. LVEF ≤45% or institutional lower limit of normal
   10. Uncontrolled hypertension (resting systolic blood pressure >180 mmHg or diastolic blood pressure >110 mmHg despite optimal medical management)
   11. Complete left or right bundle branch block
   12. Severe aortic stenosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2025-07-18 (Actual); Primary Completion 2028-06-06 (Estimated); Study Completion 2032-07-14 (Estimated)

PRIMARY OUTCOMES:
Serious Treatment Emergent Adverse Events (TEAEs) | From date of first dose to 30 days after last dose, up to 87 months
  TEAEs are defined as AEs with start or worsening date during the on-treatment period (from the first dose date of trial treatment to 30 days after the last dose date of trial treatment).

SECONDARY OUTCOMES:
TEAEs | From date of first dose to 30 days after last dose, up to 87 months
  TEAEs are defined as AEs with start or worsening date during the on-treatment period (from the first dose date of trial treatment to 30 days after the last dose date of trial treatment).
Overall Survival (OS) | From date of randomization to death from any cause, up to 87 months
  OS is defined as the time from randomization until death from any cause.
Relapse-free Survival (RFS) | From date of randomization to documented relapse or death from any cause, whichever comes first, up to 87 months
  RFS is defined as the time from randomization until documented relapse or death from any cause, whichever comes first

CONTACTS AND LOCATIONS:
Locations (57):
- United States (9):
  - John Hopkins School of Medicine, Baltimore, Maryland
  - Umass Memorial Health Care Systems, Worcester, Massachusetts
  - Roswell Park Cancer Institute, Buffalo, New York
  - Weill Cornell, New York, New York
  - Westchester Medical College, Valhalla, New York
  - Clinical Research Allicance, Westbury, New York
  - Spoknwrd Clinical Trials Inc., Easton, Pennsylvania
  - The Methodist Hospital Research Institute, Houston, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- Australia (7):
  - Royal Adelaide Hospital, Adelaide
  - Austin Health, Australia
  - St. Vincent's Hospital Melbourne, Darlinghurst
  - The Alfred Hospital, Melbourne
  - Royal Perth Hospital, Perth
  - Gold Coast University Hospital, Southport
  - Westmead Hospital, Sydney
- Brazil (8):
  - Hospital Erasto Gaertner - Liga Paranaense de Combate ao Cancer, Curitiba
  - Cetus Hospital Dia Oncologia, Minas Gerai
  - Hospital de Clínicas de Porto Alegre, Porto Alegre
  - Irmandade da Santa Casa de Misericórdia de Porto Alegre Centro Multidisciplinar de Pesquisa, Porto Alegre
  - INCA - Instituto Nacional de Câncer, Rio de Janeiro
  - "Fundacao Faculdade Regional de Medicina de Sao Jose do Rio Preto CIP - Centro Integrado de Pesquisa", San Jose Rio Preto
  - Hospital Santa Marcelina, São Paulo
  - ICESP - Instituto do Câncer do Estado de São Paulo Octavio Frias de Oliveira, São Paulo
- China (19):
  - Peking Union Medical College Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - The First Hospital of Jilin University, Changchun
  - Guangdong Provincial People's Hospital, Guangzhou
  - Nanfang Hospital of Southern Medical University, Guangzhou
  - Sun Yat-sen University Cancer center, Guangzhou
  - The First Affiliated Hosptial of Zhejiang University School of Medicine, Hangzhou
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - Zhong Da Hospital, Southeast University, Nanjing
  - The First Affiliated Hospital of Guangxi Medical University, Nanning
  - The Affiliated Hospital of Qingdao University, Qingdao
  - Huashan Hospital, Fudan University, Shanghai
  - The First Affiliated Hospital of Soochow University, Suzhou
  - Hematology Hospital of the Chinese Academy of Medical Sciences, Tianjin
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou
  - The First Affiliated Hospital of Jiaotong University, Xi'an
  - The First Affiliated Hospital of Xiamen University, Xiamen
  - The Affiliated Hospital of Xuzhou Medical College, Xuzhou
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou
- South Korea (14):
  - Inje University Haeundae Paik Hospital, Busan
  - Pusan National University Hospital, Busan
  - Kyungpook National University Hospital, Daegu
  - Yeungnam University Hospital, Daegu
  - National Cancer Center, Goyang-si
  - Gachon University Gil Medical Center, Incheon
  - Jeonbuk National University Hospital, Jeonju
  - Seoul National University Bundang Hospital, Seongnam
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Ajou University Hospital, Suwon
  - Ulsan University Hospital, Ulsan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) on completed studies and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Completed studies that has reached a global end or completion with all data set collected and analyzed, and for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents on completed clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/